CLINICAL TRIAL: NCT05277311
Title: Efficacy and Safety of LongShengZhi Capsule on Functional Recovery After Acute Ischaemic Stroke (LONGAN): A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Efficacy and Safety of LongShengZhi Capsule on Functional Recovery After Acute Ischaemic Stroke (LONGAN)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HX-DZM-202119
Record Dates: First submitted 2022-02-08; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; LongShengZhi capsule; efficacy; safety; randomized controlled trial
MeSH Terms: conditions — Ischemic Stroke | interventions — LongShengZhi

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LongShengZhi capsule (Experimental): Experimental group
  Interventions: Drug: LongShengZhi capsule
- LongShengZhi capsule placebo (Placebo Comparator): Placebo group
  Interventions: Drug: LongShengZhi capsule placebo

INTERVENTIONS:
Drug: LongShengZhi capsule — LongShengZhi capsules, orally, 5 capsules each time, three times a day.
  Arms: LongShengZhi capsule
Drug: LongShengZhi capsule placebo — LongShengZhi capsules placebo, orally, 5 capsules each time, three times a day.
  Arms: LongShengZhi capsule placebo

SUMMARY:
The aim of the study is to determine if LongShengZhi Capsule is effective and safe in patients with ischemic stroke in comparison to placebo. This trial is a prospective, multicenter, randomized, placebo-controlled, double-blinded, parallel-group, superiority trial.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke patients within 7 days of onset
* 18 years of age or older, and gender not limited
* NIHSS score of 4 to 15

Exclusion Criteria:

* Secondary stroke caused by a tumor, traumatic brain injury, hematological disease, or other diseases with a confirmed diagnosis
* Pre-stroke mRS score of more than 1
* Known severe liver or kidney dysfunction
* Known allergies for ingredients in the investigational product
* Known bleeding diathesis or coagulation disorder
* Known medical condition likely to limit survival to less than 3 months
* Pregnant women (clinically evident) or breastfeeding women
* Participation in any investigational study in the previous 3 months
* Known dementia, uncontrolled psychiatric problems
* Any condition that could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study. The judgment is left to the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1376 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with excellent outcome | 90 days after randomization
  Excellent outcome defined as a modified Rankin scale (mRS) score ≤ 1 (scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death).

SECONDARY OUTCOMES:
Distribution of the modified Rankin scale (mRS) scores | 30 days after randomization
  Modified Rankin scale (mRS) scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death.
Distribution of the modified Rankin scale (mRS) scores | 90 days after randomization
  Modified Rankin scale (mRS) scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death.
The proportion of patients with good outcome | 30 days after randomization
  Good outcome defined as a modified Rankin scale (mRS) score ≤2(scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death).
The proportion of patients with good outcome | 90 days after randomization
  Good outcome defined as a modified Rankin scale (mRS) score ≤2(scores ranged from 0 to 6, with 0 to 1 indicating no disability, 2 to 5 indicating increasing disability, and 6 indicating death).
Changes in National Institutes of Health Stroke Scale (NIHSS) scores | 90 days after randomization
  Difference of NIHSS scores (range =0-42, with higher scores indicating more severe strokes) between baseline and 30 days after randomization or 90 days after randomization.
The proportion of patients with poor quality of life | 30 days after randomization
  Poor quality of life defined as EuroQol Five Dimensions Questionnaire (EQ-D5) index score ≤0.5. The EQ-5D index score is measured on a scale of 0 (death) to 1 (full health).
The proportion of patients with poor quality of life | 90 days after randomization
  Poor quality of life defined as EuroQol Five Dimensions Questionnaire (EQ-D5) index score ≤0.5. The EQ-5D index score is measured on a scale of 0 (death) to 1 (full health).
The proportion of patients with functional independence | 30 days after randomization
  Functional independence measured withe BI, which was a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
The proportion of patients with functional independence | 90 days after randomization
  Functional independence measured withe BI, which was a commonly used scale for measuring the activity of daily living of people. Score of 10-item scale ranges from 0 (worst) to 100 (best).
Changes in Motor function | 90 days after randomization
  Motor function, measured by the Fugl-Meyer Motor Scale (FMMS) score(range from 0-100, with lower score showing worse motor status) change from baseline to 90 days after randomization.
Changes in Cognitive function | 90 days after randomization
  Cognitive function, as measured using the Montreal Cognitive Assessment (MoCA) score (range from 0 to 30, with less than 26 indicating cognitive impairment) change from baseline to 90 days after randomization.
The proportion of adverse events (AEs) | 90 days after randomization
  The proportion of AEs during the treatment.